CLINICAL TRIAL: NCT01424397
Title: A Randomized, Double-blind, Placebo Controlled, Incomplete Block, 3 Way Cross Over Study in Subjects With Allergic Rhinitis to Assess the Effect of Intranasal Repeat Doses of SB-705498 When Administered Alone or in Conjunction With Intranasal Fluticasone Propionate on the Symptoms of Rhinitis in the Vienna Allergen Challenge Chamber
Brief Title: Intranasal SB-705498 in Allergic Rhinitis (AR) Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 111924; 2011-000115-11 (EudraCT Number)
Record Dates: First submitted 2011-08-18; First posted 2011-08-29 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-08

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — SB 705498

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SB-705498 (Experimental): Experimental
  Interventions: Drug: SB-705498
- Fluticasone Propionate (Active Comparator): Active Comparator
  Interventions: Drug: FP
- Placebo (Placebo Comparator): Placebo Comparator
  Interventions: Drug: placebo
- SB-705498+FP (Experimental): Experimental
  Interventions: Drug: SB-705498; Drug: FP

INTERVENTIONS:
Drug: SB-705498 — 12mg intranasal
  Arms: SB-705498; SB-705498+FP
Drug: FP — 200ug intranasal
  Arms: Fluticasone Propionate; SB-705498+FP
Drug: placebo — placebo intranasal
  Arms: Placebo

SUMMARY:
This study is designed to look at the affect of SB-705498 on allergic rhinitis symptoms induced by an allergen chamber challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AR, as determined by the presence of rhinitis symptoms that last for several months per year, for more than 1 year and are not attributed to allergy, infections or nasal abnormalities.
2. TNSS score of >=4 following screening allergen challenge chamber.
3. Positive skin prick test for seasonal pollen
4. Positive RAST for seasonal pollen
5. Healthy as determined by responsible physician with the exception of mild asthma and AR
6. Male or female between 18 and 65 years of age inclusive.
7. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a \documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory].
   * Child-bearing potential and agrees to use one of the contraception methods listed as instructed. Female subjects must agree to use contraception until 84 days post-last treatment administration.
8. Male subjects with female partners of child-bearing potential must agree to use one contraception as instructed. This must be followed from the time of the first dose of study medication until 84 days post-last treatment administration.
9. Body weight ≥ 50 kg (males) and ≥45kg (females) and BMI within the range 19 - 29.9 kg/m2 (inclusive).
10. Screening pre-challenge FEV1 greater than or equal to 80% and baselines FEV1/FVC greater than or equal to 70% of predicted value.
11. Capable of giving written informed consent.
12. Average QTcB, < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.
13. AST and ALT < 2xULN; alkaline phosphatase and bilirubin less than or equal to 1.5xULN

Exclusion Criteria:

1. Nasal abnormalities likely to affect the outcome of the study,
2. History of frequent nosebleeds.
3. Respiratory disease other than mild asthma
4. A positive pre-study Hepatitis B or Hepatitis C result within 3 months of screening
5. Current or chronic history of liver disease, or known hepatic or biliary abnormalities
6. Positive pre-study drug/alcohol/smoking screen.
7. A positive test for HIV antibody.
8. History of regular alcohol consumption within 6 months of the study defined as:

   • An average weekly intake of >14 drinks for males or >7 drinks for females.
9. The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product prior to D1.
10. Exposure to more than four new chemical entities within 12 months prior to D1.
11. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements within 7 days prior to the first dose of study medication.
12. History of sensitivity to any of the study medications, or components
13. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
14. Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
15. Lactating females.
16. Subject is mentally or legally incapacitated.
17. Urine cotinine levels indicative of smoking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-04-14 (Actual); Primary Completion 2011-07-07 (Actual); Study Completion 2011-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bareille P, Murdoch RD, Denyer J, Bentley J, Smart K, Yarnall K, Zieglmayer P, Zieglmayer R, Lemell P, Horak F. The effects of a TRPV1 antagonist, SB-705498, in the treatment of seasonal allergic rhinitis. Int J Clin Pharmacol Ther. 2013 Jul;51(7):576-84. doi: 10.5414/CP201890. PMID 23735181
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111924 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 70 male and female participants with a history of allergic rhinitis (AR) were enrolled in this study. Study period was 14 April 2011 to 07 July 2011.
Pre-assignment Details: There were 3 study treatment periods each lasting 8 days separated by a washout of 14-20 days. Participants were randomized to 12 different sequences.
Groups:
- Treatment A First, Then B, Then D: Eligible participants received Placebo alone (treatment A) in period-1 (4 actuations per nostril of placebo matching SB-705498 alone were administered once-daily (OD) in morning for 8 days and 4 actuations per nostril of placebo matching Fluticasone propionate (FP) alone were administered OD in evening for 7 days). Participants received FP 200 microgram (μg) alone (Treatment B) in Period-2 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received 12 milligrams (mg) SB-705498 co-administered with FP (Treatment D) in Period-3 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment B First, Then A, Then D: Eligible participants received Participants received FP 200 μg alone (Treatment B) in Period-1 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-2 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received 12 mg SB-705498 co-administered with FP (Treatment D) in Period-3 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment B, Then D, Then A: Eligible participants received FP 200 μg alone (Treatment B) in Period-1 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received 12 mg SB-705498 co-administered with FP (Treatment D) in Period-2 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-3 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days).There was a 14-20 days washout between 2 treatment periods.
- Treatment A, Then D, Then B: Eligible participants received Placebo alone (treatment A) in period-1 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received 12 mg SB-705498 co-administered with FP (Treatment D) in Period-2 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-3 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment D, Then A, Then B: Eligible participants received 12 mg SB-705498 co-administered with FP (Treatment D) in Period-1 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-2 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-3 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment D, Then B, Then A: Eligible participants received 12 mg SB-705498 co-administered with FP (Treatment D) in Period-1 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-2 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-3 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment A, Then B, Then C: Eligible participants received Placebo alone (treatment A) in period-1 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-2 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received SB-705498 12 mg alone (Treatment C) in Period-3 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment B, Then A, Then C: Eligible participants received FP 200 μg alone (Treatment B) in Period-1 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-2 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received SB-705498 12 mg alone (Treatment C) in Period-3 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment B, Then C, Then A: Eligible participants received FP 200 μg alone (Treatment B) in Period-1 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received SB-705498 12 mg alone (Treatment C) in Period-2 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-3 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment A, Then C, Then B: Eligible participants received Placebo alone (treatment A) in period-1 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received SB-705498 12 mg alone (Treatment C) in Period-2 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-3 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment C, Then A, Then B: Eligible participants received SB-705498 12 mg alone (Treatment C) in Period-1 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-2 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-3 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
- Treatment C, Then B, Then A: Eligible participants received SB-705498 12 mg alone (Treatment C) in Period-1 (4 actuations per nostril [each of 1.5mg] of 12 mg SB-705498 were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). Participants received FP 200 μg alone (Treatment B) in Period-2 (4 actuations per nostril of Placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril [each of 25μg] of FP 200 μg alone were administered OD in evening for 7 days). Participants received Placebo alone (treatment A) in period-3 (4 actuations per nostril of placebo matching SB-705498 alone were administered OD in morning for 8 days and 4 actuations per nostril of placebo matching FP alone were administered OD in evening for 7 days). There was a 14-20 days washout between 2 treatment periods.
Period: Period-1 (8 Days)
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Completed | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period-1 (14-20 Days)
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Completed | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period-2 (8 Days)
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Completed | 7 | 8 | 7 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period-2 (14-20 Days)
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 7 | 8 | 7 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Completed | 7 | 8 | 7 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period-3 (8 Days)
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A
Started | 7 | 8 | 7 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Completed | 7 | 8 | 7 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects population comprised of all participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A First, Then B, Then D | Treatment B First, Then A, Then D | Treatment B, Then D, Then A | Treatment A, Then D, Then B | Treatment D, Then A, Then B | Treatment D, Then B, Then A | Treatment A, Then B, Then C | Treatment B, Then A, Then C | Treatment B, Then C, Then A | Treatment A, Then C, Then B | Treatment C, Then A, Then B | Treatment C, Then B, Then A | Total
Number analyzed (Participants) | 7 | 8 | 8 | 8 | 8 | 8 | 4 | 4 | 4 | 3 | 4 | 4 | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.6 (5.65) | 29.6 (9.24) | 28.0 (5.07) | 28.5 (9.20) | 28.5 (6.46) | 27.8 (6.34) | 24.5 (3.11) | 32.5 (10.54) | 25.3 (1.50) | 24.0 (1.00) | 28.3 (6.29) | 26.8 (11.03) | 28.1 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 3 | 4 | 4 | 2 | 0 | 4 | 2 | 1 | 1 | 33
  Male | 3 | 6 | 2 | 5 | 4 | 4 | 2 | 4 | 0 | 1 | 3 | 3 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White(Wh)-Wh/Caucasian(Ca)/European(Eu)Heritage(H) | 7 | 8 | 8 | 7 | 7 | 7 | 4 | 4 | 4 | 3 | 4 | 4 | 67
  American Indian or Alaskan Native Wh-Wh/Ca/Eu H | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Wh - Arabic/North African H | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian - South East Asian H | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Nasal Symptom Score (TNSS) and Its Individual Components on Day 8
Description: Nasal symptoms (nasal congestion, rhinorrhoea, itching and sneezing) were scored on a scale from 0 to 3 where 0= absent symptoms, 3 = severe symptoms. TNSS was calculated as the sum of the response for all 4 individual nasal symptom scores. TNSS ranged from 0 to 12, where 0=absent symptoms, 3=severe symptoms. Higher the score, more severe the symptoms. Weighted mean (WM) of TNSS and its individual components (nasal congestion, rhinorrhoea, itching and sneezing) are presented on Day 8. Weighted mean was calculated over the time interval 0 to 4 hours after start of allergen chamber challenge by calculating the area under the curve of TNSS/component from time of the first observation to time of the last observation (AUC [tf-t1 hours]) using the trapezoidal rule, and then dividing by the actual relevant time interval (tf-t1) required by participant to complete the chamber challenge assessments. A Bayesian analysis was conducted to derive the posterior probability for TNSS.
Time Frame: Day 8 of each treatment period
Population: All subjects population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Placebo: Participants administered matching placebo for SB-705498 once-daily in the form of Intranasal suspension four actuations in each nostril for 8 days in morning using Device A and matching placebo for FP once-daily in the form of Intranasal spray four actuations in each nostril in evening for 7 days using Device B.
- FP 200 μg: Participants administered matching placebo for SB-705498 once-daily in the form of Intranasal suspension four actuations in each nostril for 8 days in morning using Device A and FP 200 μg once-daily in the form of Intranasal spray four actuations in each nostril in evening for 7 days using Device B. Each spray of FP delivered approximately 25μg per actuation.
- SB-705498 12 mg: Participants administered SB-705498 12 mg once-daily in the form of Intranasal suspension four actuations in each nostril for 8 days in morning using Device A and matching placebo for FP once-daily in the form of Intranasal spray four actuations in each nostril in evening for 7 days using Device B.
- SB-705498 + FP 12 mg: Participants received SB-705498 12 mg once-daily in the form of Intranasal suspension four actuations in each nostril for 8 days in morning using Device A and FP 200 μg once-daily in the form of Intranasal spray four actuations in each nostril in evening for 7 days using Device B.
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
Score on scale
  TNSS WM | 6.53 (2.300) | 3.65 (2.360) | 6.57 (2.418) | 4.14 (2.243)
  Nasal congestion scoreWM | 1.80 (0.653) | 1.15 (0.792) | 1.82 (0.648) | 1.18 (0.715)
  Rhinorrhoea score WM | 1.67 (0.693) | 0.94 (0.726) | 1.75 (0.697) | 1.05 (0.687)
  Nasal itching score WM | 1.67 (0.760) | 0.94 (0.708) | 1.57 (0.886) | 1.17 (0.699)
  Sneezing score WM | 1.39 (0.763) | 0.62 (0.573) | 1.43 (0.785) | 0.74 (0.560)
Statistical Analysis 1: Comparison: Placebo vs FP 200 μg; Test type: Superiority or Other; Bayesian analysis: The posterior probability of a reduction in TNSS with FP alone compared to Placebo using Mixed Models Analysis was 1.0000
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Test type: Superiority or Other; Bayesian analysis: The posterior probability of a reduction in TNSS with SB-705498 alone compared to Placebo using Mixed Models Analysis was 0.7127
Statistical Analysis 3: Comparison: Placebo vs SB-705498 + FP 12 mg; Test type: Superiority or Other; Bayesian analysis: The posterior probability of a reduction in TNSS with SB-705498 + FP compared to Placebo using Mixed Models Analysis was 1.0000
Statistical Analysis 4: Comparison: FP 200 μg vs SB-705498 + FP 12 mg; Test type: Superiority or Other; Bayesian analysis: The posterior probability of a reduction in TNSS with SB-705498 + FP compared to FP alone using Mixed Models Analysis was 0.0160

2. Secondary Outcome: Mean TNSS and Its Individual Components From Day 4 to Day 8
Description: Nasal symptoms (nasal congestion, rhinorrhoea, itching and sneezing) were scored on a scale from 0 to 3 where 0= absent symptoms, 3 = severe symptoms. TNSS was calculated as the sum of the response for all 4 individual nasal symptom scores. TNSS ranged from 0 to 12, where 0=absent symptoms, 3=severe symptoms. Higher the score, more severe the symptoms. Mean of TNSS and its individual components is presented pre-evening (pm) dose on Days 4, 5, 6, 7 and pre-challenge [1 hour (hr)] on Day 8.
Time Frame: pre-evening (pm) dose on Days 4, 5, 6, 7 and pre-challenge [1 hour (hr)] on Day 8 of each treatment period
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 47
Score on a scale
  TNSS,Day 4, pre-pm dose | 3.6 (2.47) | 2.4 (2.20) | 3.3 (2.65) | 2.6 (1.94)
  TNSS,Day 5, pre-pm dose | 3.6 (2.58) | 2.0 (2.24) | 2.9 (2.60) | 2.3 (2.10)
  TNSS,Day 6, pre-pm dose | 3.3 (2.45) | 1.8 (2.03) | 2.8 (2.74) | 2.0 (2.03)
  TNSS,Day 7, pre-pm dose | 3.2 (2.26) | 1.7 (1.90) | 2.2 (2.37) | 1.9 (2.12)
  TNSS,Day 8, pre-challenge (1hr): number analyzed (Participants) | 68 | 69 | 23 | 46
  TNSS,Day 8, pre-challenge (1hr) | 2.0 (1.88) | 1.3 (1.60) | 1.9 (1.52) | 1.1 (1.45)
  Nasal congestion score code,Day 4, pre-pm dose | 1.0 (0.81) | 0.8 (0.69) | 0.9 (0.95) | 0.7 (0.65)
  Nasal congestion score code,Day 5, pre-pm dose | 0.9 (0.82) | 0.7 (0.70) | 0.7 (0.88) | 0.6 (0.64)
  Nasal congestion score code,Day 6, pre-pm dose | 0.9 (0.80) | 0.7 (0.74) | 0.8 (0.83) | 0.6 (0.68)
  Nasal congestion score code,Day 7, pre-pm dose | 0.8 (0.69) | 0.6 (0.62) | 0.7 (0.82) | 0.6 (0.65)
  Nasal congestion score code,Day 8, pre-challenge: number analyzed (Participants) | 68 | 69 | 23 | 46
  Nasal congestion score code,Day 8, pre-challenge | 0.7 (0.67) | 0.6 (0.67) | 0.6 (0.59) | 0.4 (0.58)
  Rhinorrhoea score code,Day 4, pre-pm dose | 0.9 (0.71) | 0.6 (0.76) | 0.9 (0.87) | 0.5 (0.65)
  Rhinorrhoea score code,Day 5, pre-pm dose | 0.9 (0.75) | 0.5 (0.78) | 0.9 (0.90) | 0.5 (0.66)
  Rhinorrhoea score code,Day 6, pre-pm dose | 0.8 (0.73) | 0.4 (0.65) | 0.8 (0.90) | 0.6 (0.62)
  Rhinorrhoea score code,Day 7, pre-pm dose | 0.8 (0.65) | 0.4 (0.62) | 0.6 (0.78) | 0.4 (0.69)
  Rhinorrhoea score code,Day 8, pre-challenge (1hr): number analyzed (Participants) | 68 | 69 | 23 | 46
  Rhinorrhoea score code,Day 8, pre-challenge (1hr) | 0.6 (0.69) | 0.3 (0.59) | 0.6 (0.66) | 0.3 (0.50)
  Nasal itching score code,Day 4, pre-pm dose | 0.9 (0.85) | 0.5 (0.66) | 0.7 (0.71) | 0.7 (0.71)
  Nasal itching score code,Day 5, pre-pm dose | 0.8 (0.81) | 0.4 (0.63) | 0.4 (0.66) | 0.7 (0.75)
  Nasal itching score code,Day 6, pre-pm dose | 0.8 (0.84) | 0.3 (0.58) | 0.5 (0.73) | 0.5 (0.72)
  Nasal itching score code,Day 7, pre-pm dose | 0.8 (0.80) | 0.4 (0.62) | 0.3 (0.65) | 0.5 (0.72)
  Nasal itching score code,Day 8, pre-challenge (1hr: number analyzed (Participants) | 68 | 69 | 23 | 46
  Nasal itching score code,Day 8, pre-challenge (1hr | 0.5 (0.65) | 0.3 (0.60) | 0.3 (0.49) | 0.3 (0.55)
  Sneezing score code,Day 4, pre-pm dose | 0.9 (0.78) | 0.5 (0.68) | 0.9 (0.87) | 0.6 (0.68)
  Sneezing score code,Day 5, pre-pm dose | 0.9 (0.85) | 0.4 (0.67) | 0.8 (0.83) | 0.4 (0.65)
  Sneezing score code,Day 6, pre-pm dose | 0.8 (0.82) | 0.4 (0.57) | 0.7 (0.92) | 0.4 (0.68)
  Sneezing score code,Day 7, pre-pm dose | 0.8 (0.75) | 0.3 (0.55) | 0.5 (0.73) | 0.4 (0.61)
  Sneezing score code,Day 8, pre-challenge (1hr): number analyzed (Participants) | 68 | 69 | 23 | 46
  Sneezing score code,Day 8, pre-challenge (1hr) | 0.3 (0.51) | 0.1 (0.26) | 0.4 (0.58) | 0.1 (0.31)

3. Secondary Outcome: Total Nasal Airflow on Day 8 Measured Using Active Anterior Rhinomanometry (AAR)
Description: Total Nasal Airflow is calculated as the sum of the left nostril and the right nostril airflow values. AAR is a very sensitive method of assessing clinical parameters of nasal obstruction (nasal flow, nasal resistance and nasal flow increase). A participant was instructed to breathe through one nostril while a sensor in the other nostril measured the difference in pre-nasal and choanal pressure. The system was connected to a computer. Nasal flow and nasal resistance were observed at pressure levels of 75, 150 and 300 Pascal. The defined measuring range for the flow was +-1000 milliliter per second (mL/s). Weighted means for total nasal airflow Resistance was calculated by dividing the area under the curve between 1 and 4 hours (via the linear trapezoidal method) by the total duration that the participant took to complete the chamber challenge assessments.
Time Frame: Day 8
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milliliters per second (mL/s)
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 69 | 70 | 23 | 46
Milliliters per second (mL/s) | 306.99 (17.255) | 388.34 (17.207) | 299.68 (22.806) | 379.40 (18.783)
Statistical Analysis 1: Comparison: Placebo vs FP 200 μg; Placebo versus FP 200 μg,Nasal Airflow resistance Total WM,0-4 hr; Test type: Superiority or Other; Mean Difference (Net) = 81.35, 90% CI 2-sided [60.54 to 102.15], Standard Error of Mean 12.560
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Placebo versus FP 12 mg SB-705498 , Nasal Airflow resistance Total WM, 0-4 hr; Test type: Superiority or Other; Mean Difference (Net) = -7.31, 90% CI 2-sided [-39.7 to 25.05], Standard Error of Mean 19.548
Statistical Analysis 3: Comparison: Placebo vs SB-705498 + FP 12 mg; Placebo versus SB-705498 + FP 12 mg, Nasal Airflow resistance Total WM, 0-4 hr; Test type: Superiority or Other; Mean Difference (Net) = 72.40, 90% CI 2-sided [48.28 to 96.52], Standard Error of Mean 14.567
Statistical Analysis 4: Comparison: FP 200 μg vs SB-705498 + FP 12 mg; FP 200 μg versus SB-705498 + FP 12 mg, Nasal Airflow resistance Total WM, 0-4 hr; Test type: Superiority or Other; Mean Difference (Net) = -8.95, 90% CI 2-sided [-33.1 to 15.22], Standard Error of Mean 14.592

4. Secondary Outcome: Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Following Repeat Doses of SB-705498 or or SB-705498 Matching Placebo
Description: The RQLQ composed of 28 items covering 7 domains of health. Each question is scored on a scale of 0 to 6 (where, 0 = not troubled and 6 = extremely troubled). 7 domains were: Activities (3 items):1, 2, 3;Sleep (3 items): 4, 5, 6; Non-nose/eye symptoms (7 items): 7, 8, 9, 10, 11, 12, 13; Practical Problems (3 items): 14, 15, 16; Nasal Symptoms (4 items): 17, 18, 19, 20; Eye Symptoms (4 items): 21, 22, 23, 24; Emotional (4 items): 25, 26, 27, 28 consisted of total 28 items. Domain activity score = total post-baseline score for individualized activity items answered on both visits divided by total Baseline score for individualized activity items answered on both visits multiplied by the Baseline score for item(s) missing post-baseline. The global RQLQ score was calculated by averaging all 28 item scores, which ranges from 0 to 6 (where, 0 = not troubled and 6 = extremely troubled). Higher scores indicate worsening of symptoms.
Time Frame: Day 8
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 69 | 70 | 23 | 46
Score on a scale | 1.67 (0.119) | 0.99 (0.118) | 1.66 (0.177) | 1.14 (0.135)
Statistical Analysis 1: Comparison: Placebo vs FP 200 μg; Test type: Superiority or Other; Mean Difference (Net) = -0.68, 90% CI 2-sided [-0.87 to -0.49], Standard Error of Mean 0.113
Statistical Analysis 2: Comparison: Placebo vs SB-705498 12 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.01, 90% CI 2-sided [-0.30 to 0.27], Standard Error of Mean 0.173
Statistical Analysis 3: Comparison: Placebo vs SB-705498 + FP 12 mg; Test type: Superiority or Other; Mean Difference (Net) = -0.52, 90% CI 2-sided [-0.74 to -0.31], Standard Error of Mean 0.130
Statistical Analysis 4: Comparison: FP 200 μg vs SB-705498 + FP 12 mg; Test type: Superiority or Other; Mean Difference (Net) = 0.15, 90% CI 2-sided [-0.06 to 0.37], Standard Error of Mean 0.130

5. Secondary Outcome: Area Under Concentration-time Curve (AUC) for SB-705498 on Day 8
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at indicated time points of each treatment period. AUC0-t was calculated by the linear trapezoidal method. AUC0-infinity was calculated as the sum of the AUC0-t plus the ratio of the last measurable plasma concentration to the elimination rate constant, where first-order elimination or terminal rate constant was calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the last three (or more) non-zero plasma concentrations. Values were reported as Least Squares Geometric Means with respective % CV.
Time Frame: Period 1: Day 1 (post dose 1 and 5 h) and 8 (Pre-dose (0.0 h), post dose 1 and 5 h), Period 2 and 3: Day 1 (Pre-dose 0.0 h, post dose 1 and 5 h) and 8 (Pre-dose (0.0 h), post dose 1 and 5 h)
Population: The 'Pharmacokinetic Population' is defined as participants in the 'All Subjects' population for whom a pharmacokinetic sample was obtained and analyzed. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per mililiter (ng.h/mL)
Arm/Group | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 23 | 46
nanograms*hour per mililiter (ng.h/mL) | 588.26 (71.4) | 608.84 (74.2)

6. Secondary Outcome: Maximum Observed Concentration (Cmax) for SB-705498 on Day 8
Description: Plasma samples for pharmacokinetic analysis were drawn at indicated time points of each treatment period. Cmax was defined as maximal measured plasma concentration over the time span specified. Values were reported as least squares geometric means with respective geometric coefficient of variation (% CV).
Time Frame: as for outcome 5
Population: Pharmacokinetic Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per mililiter (ng/mL)
Arm/Group | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 23 | 46
nanograms per mililiter (ng/mL) | 145.958 (68.8) | 154.231 (71.0)

7. Secondary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance (PCI)
Description: Vital signs assessment included heart rate, blood pressure, and temperature. Criteria for vital sign values meeting potential clinical concern included: systolic blood pressure (SBP) <85 and >160 millimeters of mercury (mm Hg), diastolic blood pressure (DBP) < 45 and > 100 mm Hg, temperature <36 and >37.5 Degree Celsius and heart Rate <40 and >110 beats per minute. Only parameters with PCI values are reported.
Time Frame: Up to Week 16
Population: All Subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
Participants
  Temperature,Low,period 3 | 2 | 0 | 0 | 0
  Temperature,Low,Follow up | 2 | 1 | 0 | 0

8. Secondary Outcome: Change From Baseline in ECG Values: Heart Rate
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated heart rate and measured PQ, QRS, QT, and QTc intervals. Baseline was assessment on Day 1. Change from Baseline was the values at specified time points subtracted by the Baseline value.
Time Frame: Baseline and Day 8 of each treatment period
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- SB-705498 + FP 12 mg: Participants administered SB-705498 12 mg once-daily in the form of Intranasal suspension four actuations in each nostril for 8 days in morning using Device A and matching placebo for FP once-daily in the form of Intranasal spray four actuations in each nostril in evening for 7 days using Device B.
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
beats per minute (bpm) | -0.2 (11.32) | -4.7 (10.80) | -4.8 (8.09) | -2.6 (11.19)

9. Secondary Outcome: Change From Baseline in ECG Values: PR Interval, QRS Duration, QT Interval, QTcB, QTcF
Description: Single 12-lead ECGs were obtained at each time point during the study using an ECG machine that automatically calculated heart rate and measured PQ, QRS, QT, QTc corrected by Bazett's formula (QTcB) and QTc corrected by Fridericia's formula (QTcF). Baseline was assessment on Day 1. Change from Baseline was the values at specified time points subtracted by the Baseline value.
Time Frame: Baseline and Day 8 of each treatment period
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliseconds (msec)
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
Milliseconds (msec)
  PR Interval | 2.7 (8.31) | -1.2 (9.38) | 4.5 (9.29) | 0.4 (9.73)
  QRS Duration | 0.8 (6.30) | 2.2 (5.52) | 0.8 (5.92) | -0.2 (5.05)
  QT Interval | -1.5 (21.47) | 4.6 (22.12) | -0.3 (17.50) | 2.5 (17.93)
  QTcB | -3.6 (17.30) | -9.3 (18.44) | -13.9 (20.79) | -4.1 (21.10)
  QTcF | -2.9 (13.16) | -4.4 (13.37) | -9.0 (16.53) | -1.9 (13.33)

10. Secondary Outcome: Number of Participants With Hematology Parameters of PCI
Description: The PCC range for hematology parameters included white blood cell count, low: 0.67, high 1.82, neutrophil count, low: 0.83, Hemoglobin, male- high 1.03, female- high 1.13, hematocrit, male- high 1.02, female- high 1.17, Platelet Count, low: 0.67, high: 1.57, lymphocytes, low 0.81. Only parameters with PCI values are reported.
Time Frame: Up to Week 16
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
Participants
  Total Neutrophils,low | 7 | 9 | 2 | 4
  Hematocrit,high | 0 | 0 | 1 | 0
  Hemoglobin,high | 0 | 0 | 1 | 0

11. Secondary Outcome: Number of Participants With Clinical Biochemistry Parameters of PCI
Description: The PCC range for clinical chemistry parameters included albumin, low: 0.86, millimole per liter (mmol)/L, calcium, low: 0.91, high: 1.06, glucose. Low: 0.71, high: 1.41, Potassium, low: 0.86, high: 1.10, Sodium, low: 0.96, high: 1.03, Total CO2, Low: 0.86, high: 1.14, Creatinine, in male, Low: <75 micromole per liter (μmol/L), high: >110 μmol/L, female, Low: <65 μmol/L, high: >95, Blood Urea Nitrogen (BUN), high: >1.5xULN mmol/L, Uric Acid, in male, Low: < 180 μmol/L, high: > 480 μmol/L, female, Low: < 120 μmol/L, high: > 420. Only parameters with PCI values are reported.
Time Frame: Up to Week 16
Population: All subjects population. Only those participants available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
Number analyzed (Participants) | 68 | 69 | 23 | 46
Participants
  Creatinine,Low | 19 | 25 | 6 | 14
  Creatinine,High | 2 | 2 | 1 | 2
  Aspartate Amino Transferase,High | 1 | 1 | 1 | 0
  Potassium,High | 2 | 4 | 2 | 5
  Uric acid,High | 1 | 0 | 1 | 1
  Gamma Glutamyl Transferase,High | 1 | 1 | 2 | 1
  Total Bilirubin,High | 1 | 1 | 1 | 1
  Alanine Amino Transferase,High | 0 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-SAEs and SAEs were collected from start of the treatment up to Week 16.
Description: All subject population was used for collection of adverse events
Arm/Group | Placebo | FP 200 μg | SB-705498 12 mg | SB-705498 + FP 12 mg
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/69 | 0/23 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/69 | 0/23 | 0/47
Other Adverse Events (participants affected / at risk) | 24/68 | 28/69 | 13/23 | 19/47
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=68) | FP 200 μg (N=69) | SB-705498 12 mg (N=23) | SB-705498 + FP 12 mg (N=47)
Hypersensitivity (Immune system disorders) | 12 | 11 | 7 | 10
Food allergy (Immune system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 9 | 11 | 5 | 5
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1
Influenza (Infections and infestations) | 0 | 2 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.